CLINICAL TRIAL: NCT01622543
Title: A Randomized Phase II Study of Reolysin in Combination With FOLFOX6 and Bevacizumab or FOLFOX6 and Bevacizumab Alone in Patients With Metastatic Colorectal Cancer.
Brief Title: Reolysin in Combination With FOLFOX6 and Bevacizumab or FOLFOX6 and Bevacizumab Alone in Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Oncolytics Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I210
Record Dates: First submitted 2012-06-12; First posted 2012-06-19 (Estimated); Results first posted 2019-12-13 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2020-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Folfox protocol; Bevacizumab; reolysin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Folfox plus Bevacizumab and Reolysin (Active Comparator)
  Interventions: Drug: Folfox plus Bevacizumab and reolysin
- Folfox plus Bevacizumab (Active Comparator)
  Interventions: Drug: Folfox plus Bevacizumab

INTERVENTIONS:
Drug: Folfox plus Bevacizumab and reolysin — FOLFOX6/bevacizumab given every 14 days plus reolysin days 1-5 on cycles 1, 2, 4, 6, 8 and alternate cycles thereafter
  Arms: Folfox plus Bevacizumab and Reolysin
Drug: Folfox plus Bevacizumab — FOLFOX6/bevacizumab given every 14 days.
  Arms: Folfox plus Bevacizumab

SUMMARY:
The purpose of this study is to find out if giving reolysin in combination with FOLFOX6/ bevacizumab can offer better results than standard therapy with FOLFOX6/ bevacizumab.

DETAILED DESCRIPTION:
Researchers doing this study also want to evaluate the side effects of reolysin when given together with FOLFOX6/ bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histological diagnosis of colorectal adenocarcinoma.
* All patients must have a formalin fixed paraffin embedded tissue block (from their primary or metastatic tumour) available for translational studies and must have provided informed consent for the release of the block.
* Presence of clinically and/or radiologically documented disease. All radiology studies must be performed within 28 days prior to randomization (within 35 days if negative). All patients must have measurable disease as defined by RECIST 1.1.

The criteria for defining measurable disease are as follows:

Chest X-ray ≥ 20 mm CT/MRI scan (with slice thickness of < 5 mm) ≥ 10 mm longest diameter Physical exam (using calipers) ≥ 10 mm Lymph nodes by CT scan ≥ 15 mm measured in short axis

* Patients must have advanced and or metastatic disease, for which no curative therapy exists and for which systemic therapy is indicated.
* ECOG performance of 0, 1 or 2.
* Age ≥ 18 years of age.
* Previous Therapy

Surgery:

Previous major surgery is permitted provided that it has been at least 21days prior to patient randomization and that wound healing has occurred.

Chemotherapy:

Patients may NOT have received any prior cytotoxic chemotherapy for advanced or metastatic disease. Prior adjuvant fluoropyrimidine-based therapy is permitted provided completed at least one year prior to enrollment and the regimen did not include oxaliplatin or bevacizumab. Exceptions may be made for low dose chemotherapy given as a radiosensitizing agent.

Other Therapy:

Patients may have received other therapies including immunotherapy, or with signal transduction inhibitors, providing that the patient has recovered from all reversible drug related toxicity (with the exception of alopecia) and adequate washout period has been met.

Radiation:

Prior external beam radiation is permitted provided a minimum of 4 weeks has elapsed between the last dose and enrollment to the trial. Exceptions may be made for low dose, non-myelosuppressive radiotherapy after consultation with NCIC CTG.

* Laboratory Requirements (must be done within 7 days prior to randomization)

Hematology:

Granulocytes (AGC) ≥ 1.5 x 10^9/L Platelets ≥ 100 x 10^9/L

Biochemistry:

Serum creatinine ≤ 1.5 x ULN Total bilirubin ≤ 1.0 x ULN (unless elevated secondary to conditions such as Gilbert's disease) ALT and AST ≤ 3 x ULN (Note: ≤ 5 x ULN if documented liver metastasis) Proteinuria < 2g/24 hrs (screen using spot testing; if ≥ grade 2 repeat with mid-stream urine - if still ≥ grade 2 then urine collection for 24 hours to confirm <2g/24hrs)

* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate.

Patients who cannot give informed consent (i.e. mentally incompetent patients, or those physically incapacitated such as comatose patients) are not to be recruited into the study. Patients competent but physically unable to sign the consent form may have the document signed by their nearest relative or legal guardian. Each patient will be provided with a full explanation of the study before consent is requested.

* Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: 2 hour's driving distance) placed on patients being considered for this trial. Investigators must assure themselves that the patients registered on this trial will be available for complete documentation of the treatment, adverse events, response assessment and follow-up.
* Patient is able (i.e. sufficiently fluent) and willing to complete the quality of life (EORTC QLQ-C30) in either English or French. The baseline assessment must already have been completed. Inability (illiteracy in English or French, loss of sight, or other equivalent reason) to complete the questionnaires will not make the patient ineligible for the study. However, ability but unwillingness to complete the questionnaires will make the patient ineligible. The baseline assessment must be completed within 14 days prior to randomization.
* In accordance with NCIC CTG policy, protocol treatment is to begin within 5 working days of patient randomization.

Exclusion Criteria:

* Patients with a history of other malignancies, except for adequately treated non-melanoma skin cancer or solid tumours curatively treated with no evidence of disease for ≥ 3 years. (Please call NCIC CTG if any questions about the interpretation of this criterion).
* Patients who are on immunosuppressive therapy or have known HIV infection or active hepatitis B or C.
* Patients with active or uncontrolled infections or with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol.
* Patients with significant cardiac (including uncontrolled hypertension) or pulmonary disease, or active CNS disease or infection.
* Patients are not eligible if they have a known hypersensitivity to the study drug(s) or their components.
* Patients with history of central nervous system metastases or untreated spinal cord compression.
* Patients who have had prior treatment with oxaliplatin or bevacizumab, who have contraindications to treatment with 5FU (for e.g. known DPD deficiency or severe cardiac disease), and or neuropathy > grade 1.
* Patients who are not sterile unless they use an adequate method of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2012-10-26 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2018-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Jonker, Study Chair — Ottawa Health Research Institute - General Division; Patricia Tang, Study Chair — Tom Baker Cancer Centre, Calgary, Canada
Locations (10):
- Canada (10):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - McGill University - Dept. Oncology, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jonker DJ, Tang PA, Kennecke H, Welch SA, Cripps MC, Asmis T, Chalchal H, Tomiak A, Lim H, Ko YJ, Chen EX, Alcindor T, Goffin JR, Korpanty GJ, Feilotter H, Tsao MS, Theis A, Tu D, Seymour L. A Randomized Phase II Study of FOLFOX6/Bevacizumab With or Without Pelareorep in Patients With Metastatic Colorectal Cancer: IND.210, a Canadian Cancer Trials Group Trial. Clin Colorectal Cancer. 2018 Sep;17(3):231-239.e7. doi: 10.1016/j.clcc.2018.03.001. Epub 2018 Mar 8. PMID 29653857
- [Derived] Provencher DM, Gallagher CJ, Parulekar WR, Ledermann JA, Armstrong DK, Brundage M, Gourley C, Romero I, Gonzalez-Martin A, Feeney M, Bessette P, Hall M, Weberpals JI, Hall G, Lau SK, Gauthier P, Fung-Kee-Fung M, Eisenhauer EA, Winch C, Tu D, MacKay HJ. OV21/PETROC: a randomized Gynecologic Cancer Intergroup phase II study of intraperitoneal versus intravenous chemotherapy following neoadjuvant chemotherapy and optimal debulking surgery in epithelial ovarian cancer. Ann Oncol. 2018 Feb 1;29(2):431-438. doi: 10.1093/annonc/mdx754. PMID 29186319

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 patients were enrolled in a safety run-in phase of the study before randomized component was started. These 6 patients were not included in the final analysis.
Groups:
- Folfox Plus Bevacizumab and Reolysin: Folfox plus Bevacizumab and reolysin: FOLFOX6/bevacizumab infusion on day 1 of a 14 day cycle (IV bevacizumab 5mg/kg over 1 hour, oxaliplatin 85mg/m^2 and leucovorin 400 mg/m^2 concurrently over 2 hours, bolus fluorouracil 400 mg/m^2 after leucovorin, and continuous infusion of fluorouracil 2400 mg/m^2 over 46 hours) and reolysin 3x10^10 TCID_50 over 1 hour on days 1-5 of cycle 2, 4, 6, 8 and alternate cycles thereafter.
- Folfox Plus Bevacizumab: Folfox plus Bevacizumab: FOLFOX6/bevacizumab infusion on day 1 of a 14 day cycle (IV bevacizumab 5mg/kg over 1 hour, oxaliplatin 85mg/m^2 and leucovorin 400 mg/m^2 concurrently over 2 hours, bolus fluorouracil 400 mg/m^2 after leucovorin, and continuous infusion of fluorouracil 2400 mg/m^2 over 46 hours).
Period: Overall Study
Arm/Group | Folfox Plus Bevacizumab and Reolysin | Folfox Plus Bevacizumab
Started | 51 | 52
Completed | 51 | 52
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients randomized to this study
Groups:
- Total: Total of all reporting groups
Arm/Group | Folfox Plus Bevacizumab and Reolysin | Folfox Plus Bevacizumab | Total
Number analyzed (Participants) | 51 | 52 | 103
Age, Continuous [Median (Full Range); unit: years] | 60 [34 to 79] | 59 [31 to 78] | 60 [31 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 40
  Male | 32 | 31 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 51 | 51 | 102
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 51 | 52 | 103
ECOG Performance Status [Count of Participants; unit: Participants] — 0: Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair
  5. Dead
  Participants
    0 | 20 | 27 | 47
    1 | 29 | 23 | 52
    2 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Time from the day of randomization until the first observation of objective disease relapse or progression, or the appearance of new lesions or death due to any cause. If a patient had not relapsed/progressed or died, PFS was censored on the date of last disease assessment defined as the earliest test date of target lesion or non-target lesions (if patient had no target lesions). Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 19 months
Population: All patients randomized
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Folfox Plus Bevacizumab and Reolysin | Folfox Plus Bevacizumab
Number analyzed (Participants) | 51 | 52
Months | 7.33 [5.42 to 9.17] | 9.13 [7.39 to 11.83]
Statistical Analysis 1: Comparison: Folfox Plus Bevacizumab and Reolysin vs Folfox Plus Bevacizumab; Test type: Superiority; p = 0.046, Log Rank; Hazard Ratio (HR) = 1.59, 95% CI 2-sided [1.00 to 2.53]

2. Secondary Outcome: Changes in CEA Levels
Description: Changes in CEA level from baseline to week 28 during treatment.
Time Frame: Baseline and at 28 weeks
Population: All patients who had CEA levels measures at baseline and week 28.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Folfox Plus Bevacizumab and Reolysin | Folfox Plus Bevacizumab
Number analyzed (Participants) | 18 | 20
ng/mL | -14209.4 (58829.51) | -1107.99 (2670.55)
Statistical Analysis 1: Comparison: Folfox Plus Bevacizumab and Reolysin vs Folfox Plus Bevacizumab; Test type: Superiority; p = 0.45, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Objective Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response Rate =Proportion of (CR + PR) observed over all randomized patients.
Time Frame: 19 months
Population: All patients randomized to this study
Measure: Count of Participants; unit: Participants
Arm/Group | Folfox Plus Bevacizumab and Reolysin | Folfox Plus Bevacizumab
Number analyzed (Participants) | 51 | 52
Participants | 27 | 18
Statistical Analysis 1: Comparison: Folfox Plus Bevacizumab and Reolysin vs Folfox Plus Bevacizumab; Test type: Superiority; p = 0.06, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.09, 95% CI 2-sided [0.96 to 4.55]

4. Secondary Outcome: Overall Survival
Description: Time from randomization to death from any cause or censored at the time of last known alive
Time Frame: From date of randomization to death from any cause or censored at the time of last known alive, assessed up to 49 months
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Folfox Plus Bevacizumab and Reolysin | Folfox Plus Bevacizumab
Number analyzed (Participants) | 51 | 52
Months | 19.3 [14.4 to 23.3] | 20.0 [14.5 to 26.0]
Statistical Analysis 1: Comparison: Folfox Plus Bevacizumab and Reolysin vs Folfox Plus Bevacizumab; Test type: Superiority; p = 0.36, Log Rank; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [0.78 to 1.98]

ADVERSE EVENTS:
Time Frame: A median follow-up of 33.5 months
Arm/Group | Folfox Plus Bevacizumab and Reolysin | Folfox Plus Bevacizumab
All-Cause Mortality (participants affected / at risk) | 39/51 | 39/52
Serious Adverse Events (participants affected / at risk) | 22/51 | 18/52
Other Adverse Events (participants affected / at risk) | 51/51 | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Folfox Plus Bevacizumab and Reolysin (N=51) | Folfox Plus Bevacizumab (N=52)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 4
Acute coronary syndrome (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0
Heart failure (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Colonic fistula (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 2 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Oral hemorrhage (Gastrointestinal disorders) | 0 | 1
Other gastrointestinal disorders (Gastrointestinal disorders) | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal obstruction (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2
Fatigue (General disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 4 | 0
Other infections and infestations (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Prolapse of intestinal stoma (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Other neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 1 | 1
Stroke (Nervous system disorders) | 1 | 0
Transient ischemic attacks (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Folfox Plus Bevacizumab and Reolysin (N=51) | Folfox Plus Bevacizumab (N=52)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 5
Sinus tachycardia (Cardiac disorders) | 2 | 3
Blurred vision (Eye disorders) | 4 | 5
Dry eye (Eye disorders) | 4 | 2
Watering eyes (Eye disorders) | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 27 | 35
Bloating (Gastrointestinal disorders) | 2 | 4
Colonic perforation (Gastrointestinal disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 37 | 32
Diarrhea (Gastrointestinal disorders) | 35 | 36
Dry mouth (Gastrointestinal disorders) | 6 | 4
Dyspepsia (Gastrointestinal disorders) | 10 | 12
Flatulence (Gastrointestinal disorders) | 7 | 9
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 | 8
Hemorrhoids (Gastrointestinal disorders) | 8 | 2
Mucositis oral (Gastrointestinal disorders) | 27 | 31
Nausea (Gastrointestinal disorders) | 36 | 34
Oral hemorrhage (Gastrointestinal disorders) | 1 | 4
Oral pain (Gastrointestinal disorders) | 4 | 1
Other gastrointestinal disorders (Gastrointestinal disorders) | 2 | 5
Rectal hemorrhage (Gastrointestinal disorders) | 9 | 8
Rectal pain (Gastrointestinal disorders) | 5 | 7
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 1
Toothache (Gastrointestinal disorders) | 5 | 1
Vomiting (Gastrointestinal disorders) | 24 | 22
Chills (General disorders) | 24 | 11
Edema face (General disorders) | 3 | 1
Edema limbs (General disorders) | 18 | 10
Fatigue (General disorders) | 45 | 51
Fever (General disorders) | 31 | 15
Flu like symptoms (General disorders) | 4 | 5
Infusion related reaction (General disorders) | 2 | 5
Malaise (General disorders) | 2 | 3
Non-cardiac chest pain (General disorders) | 7 | 4
Pain (General disorders) | 6 | 9
Allergic reaction (Immune system disorders) | 0 | 4
Gum infection (Infections and infestations) | 0 | 3
Lung infection (Infections and infestations) | 6 | 1
Other infections and infestations (Infections and infestations) | 0 | 3
Sepsis (Infections and infestations) | 4 | 1
Sinusitis (Infections and infestations) | 3 | 2
Skin infection (Infections and infestations) | 2 | 5
Upper respiratory infection (Infections and infestations) | 8 | 12
Urinary tract infection (Infections and infestations) | 4 | 2
Bruising (Injury, poisoning and procedural complications) | 3 | 5
Anorexia (Metabolism and nutrition disorders) | 38 | 36
Dehydration (Metabolism and nutrition disorders) | 5 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 18
Chest wall pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 15
Dizziness (Nervous system disorders) | 6 | 6
Dysesthesia (Nervous system disorders) | 5 | 5
Dysgeusia (Nervous system disorders) | 15 | 21
Headache (Nervous system disorders) | 23 | 24
Memory impairment (Nervous system disorders) | 5 | 1
Paresthesia (Nervous system disorders) | 5 | 7
Peripheral motor neuropathy (Nervous system disorders) | 0 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 45 | 47
Syncope (Nervous system disorders) | 3 | 0
Tremor (Nervous system disorders) | 4 | 1
Anxiety (Psychiatric disorders) | 6 | 12
Depression (Psychiatric disorders) | 3 | 5
Insomnia (Psychiatric disorders) | 19 | 24
Acute kidney injury (Renal and urinary disorders) | 4 | 0
Hematuria (Renal and urinary disorders) | 3 | 3
Proteinuria (Renal and urinary disorders) | 7 | 5
Urinary frequency (Renal and urinary disorders) | 4 | 2
Pelvic pain (Reproductive system and breast disorders) | 2 | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 11 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 25
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 21 | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 24 | 28
Hiccups (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Other respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 12 | 4
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 25 | 20
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 11
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 | 4
Nail discoloration (Skin and subcutaneous tissue disorders) | 3 | 4
Other skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 6 | 5
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 4
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 6
Periorbital edema (Skin and subcutaneous tissue disorders) | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 5
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 5
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 6 | 14
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 3
Flushing (Vascular disorders) | 1 | 5
Hematoma (Vascular disorders) | 3 | 2
Hot flashes (Vascular disorders) | 3 | 1
Hypertension (Vascular disorders) | 19 | 11
Hypotension (Vascular disorders) | 4 | 2
Thromboembolic event (Vascular disorders) | 14 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-12-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT01622543/Prot_000.pdf
  • Statistical Analysis Plan (2015-03-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT01622543/SAP_001.pdf